CLINICAL TRIAL: NCT02595762
Title: A Disease Registry Study to Prospectively Observe Treatment Patterns and Outcomes in Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Treatment Patterns and Outcomes in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28801
Record Dates: First submitted 2015-10-28; First posted 2015-11-03 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants With HER2-Positive Breast Cancer: Enrolled participants will receive treatment and clinical assessments for their HER2-positive unresectable LABC/MBC as determined by their treating physician, according to the standard of care and routine clinical practice at each site. Participants will be followed until death, withdrawal of consent or study termination, whichever occurs first. Study protocol does not specify any particular drug or treatment regimen.

SUMMARY:
This disease registry is a prospective, multicenter non-interventional study designed to observe anti-cancer treatment regimens and clinical outcomes in participants with HER2-positive unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HER2-positive unresectable LABC or MBC within 6 months prior to enrollment

Exclusion Criteria:

* None specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disease registry data will be collected among participants with HER2-positive unresectable LABC or MBC.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Each Unique Treatment Regimen Overall | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Unique Treatment Regimen as First-Line Versus Subsequent-Line Therapy | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Unique Treatment Regimen Sequence | Baseline up to approximately 8 years
Progression-Free Survival (PFS) | From start date of anti-cancer treatment regimen to the date of either disease progression or death (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-/country-specific medical practice. Study protocol does not specify any particular method of assessment.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Treatment Regimen, by Participant Characteristics | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Treatment Regimen, by Country/Region | Baseline up to approximately 8 years
Overall Survival (OS) | From the date of initiation of treatment to the date of death from any cause (up to approximately 8 years)
Number of Treatment Regimens Received | Baseline up to approximately 8 years
Percentage of Participants With Complete Response (CR) or Partial Response (PR) - Objective Response Rate (ORR) | From the date of initiation of treatment to the date of disease progression or death from any cause (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-/country-specific medical practice. Study protocol does not specify any particular method of assessment.
Duration of Response (DOR) | From date of first response (CR or PR) to the date of disease progression (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-/country-specific medical practice. Study protocol does not specify any particular method of assessment.
Percentage of Participants by Reasons for Treatment Modification | Baseline up to approximately 8 years
EuroQoL 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Score | Baseline up to approximately 8 years
Functional Assessment of Cancer Therapy-Breast (FACT-B) Questionnaire Score | Baseline up to approximately 8 years
Work Productivity and Activity Impairment-General Health (WPAI-GH) Questionnaire Score | Baseline up to approximately 8 years
Percentage of Participants With HER2 Retesting | Baseline up to approximately 8 years
Percentage of Participants With HER2 Overexpression, as Assessed Using In Situ Hybridization or Immunohistochemistry | Baseline up to approximately 8 years
Healthcare Resource Utilization - Total Healthcare Cost | Baseline up to approximately 8 years
Healthcare Resource Utilization - Percentage of Participants Who Are Hospitalized | Baseline up to approximately 8 years
Healthcare Resource Utilization - Length of Hospitalization | Baseline up to approximately 8 years
Healthcare Resource Utilization - Percentage of Participants With Emergency Room Visit | Baseline up to approximately 8 years
Healthcare Resource Utilization - Percentage of Participants With Outpatient Visit | Baseline up to approximately 8 years
Healthcare Resource Utilization - Cost of Disease Related Out-of-Pocket Healthcare Expenditures | Baseline up to approximately 8 years
Healthcare Resource Utilization - Indirect Disease Related Cost | Baseline up to approximately 8 years
Healthcare Resource Utilization - Number of Working Hours Missed Among Informal Caregivers due to Disease-Related Caregiving Responsibilities | Baseline up to approximately 8 years
Healthcare Resource Utilization - Percentage of Participants Receiving Monetary Social Benefits | Baseline up to approximately 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Bank of Cyprus Oncology Center, Nicosia, Cyprus
- Greece (11):
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - Anticancer Hospital Ag. Savas ; 2Nd Dept. of Oncology - Internal Medicine, Athens
  - ARETAIEION UNIVERSITY HOSPITAL; oncology unit, Athens
  - 251 Air Force General Hospital-Oncology Clinic, Athens
  - Agioi Anargyroi; 3Rd Dept. of Medical Oncology, Athens
  - IASO, Athens
  - IASO General Hospital of Athens, Athens
  - Attikon University Hospital; 4th Department of Internal Medicine, Haidari
  - Metropolitan Hospital; 2Nd Oncology Clinic, Piraeus
  - Theagenio Anticancer Hospital; 3Rd Oncology Clinic, Thessaloniki
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki